CLINICAL TRIAL: NCT03710317
Title: Carbetocin Versus Buccal Misoprostol Plus IV Tranexamic Acid for Prevention of Postpartum Hemorrhage at Cesarean Section: A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Carbetocin Versus Buccal Misoprostol Plus IV Tranexamic Acid for Prevention of Postpartum Hemorrhage at Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: aswu/274/7/18
Record Dates: First submitted 2018-10-13; First posted 2018-10-18 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; postpartum hemorrhage; buccal misoprostol; carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Tranexamic Acid; Misoprostol

STUDY DESIGN:
Intervention Model Description: Study drug administration Group 1 100 μg carbetocin ampoule will be diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby
  Group 2 400 μg buccal misoprostol (2 tablets of 200 μg) will be given after spinal anesthesia and few minutes before skin incision in addition to 1 gm tranexamic acid in 100 mL of intravenous solution infusion over 15 min.
Who Masked: Participant, Care Provider, Investigator
Masking Description: a double-blinded randomized placebo-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbetocin (Active Comparator): 100 μg carbetocin ampoule will be diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby
  Interventions: Drug: carbetocin
- Tranexamic acid plus misoprostol (Experimental): 400 μg buccal misoprostol (2 tablets of 200 μg) will be given after spinal anesthesia and few minutes before skin incision in addition to 1 gm tranexamic acid in 100 mL of intravenous solution infusion over 15 min.
  Interventions: Drug: Tranexamic Acid; Drug: misoprostol

INTERVENTIONS:
Drug: carbetocin — 100 μg carbetocin ampoule will be diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby
  Other Names: Active Comparator
  Arms: carbetocin
Drug: Tranexamic Acid — 1 gm tranexamic acid in 100 mL of intravenous solution infusion over 15 min.
  Other Names: Experimental
  Arms: Tranexamic acid plus misoprostol
Drug: misoprostol — Group 2 400 μg buccal misoprostol (2 tablets of 200 μg) will be given after spinal anesthesia and few minutes before skin incision
  Other Names: expremental
  Arms: Tranexamic acid plus misoprostol

SUMMARY:
The Millennium Development Goal of reducing the maternal mortality ratio by 75 % by 2015 will remain beyond our reach unless we prioritize the prevention and treatment of postpartum hemorrhage(PPH) in low-resource countries. Consequently, the administration of uterotonic drugs during cesarean section (CS) and in the third stage of labor for vaginal delivery has become essential to diminish the risk of PPH and improve maternal safety.

Oxytocin is regarded as the gold standard uterotonic agent but only has a half-life of 4-10 min; therefore, at cesarean section oxytocin must be administered as a continuous intravenous infusion to attain sustained uterotonic activity throughout the surgical procedure and immediate postpartum period.

Misoprostol is a prostaglandin E1 analog proven in several randomized controlled trials to be effective in preventing PPH because of its strong uterotonic effects. In addition, misoprostol is inexpensive, stable at room temperature, and easy to administer.

Misoprostol has been broadly studied in the prevention and treatment of PPH after vaginal delivery; however, its use in conjunction with CS has not been investigated as much.

The buccal route is recognized as having the greatest benefit due to its rapid uptake, long-acting effect, and greatest bioavailability compared with other routes of misoprostol administration.

Carbetocin is a long-acting synthetic analog of oxytocin that can be administered as a single-dose injection; intravenously administered carbetocin has a half-life of approximately 40 min.

A single intravenous bolus of carbetocin produces a tetanic uterine contraction within 2 min and persists for an average of 60 min following injection.

The aim of this study was to compare the effectiveness of combined buccal misoprostol and IV tranexamic acid (TA)with intravenous carbetocin for prevention of PPH in patients with risk factors during cesarean section.

DETAILED DESCRIPTION:
Eligible and consenting participants were randomized via a computer-generated random number sequence into one of two groups: one group received a pre-prepared sealed and opaque packet containing 400 μg of misoprostol (2 tablets of 200 μg), 2 ampoules of TA. The other group received similar packets containing two placebo tablets, two placebo ampoules (distilled water) and separate carbetocin ampoule (100 μg) for slow intravenous injection. The misoprostol and placebo tablets were similar in size, shape, and color, and ampoules of TA and carbetocin will be also similar to placebo. Randomization was done by the resident doctors immediately before transfer to the theater, whereas preparation of packets and confidential record maintenance was done by the labor room nursing staff.

Study drug administration Group 1 100 μg carbetocin ampoule will be diluted in 10 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist after the birth of the baby

Group 2 400 μg buccal misoprostol (2 tablets of 200 μg) will be given after spinal anesthesia and few minutes before skin incision in addition to 1 gm tranexamic acid in 100 mL of intravenous solution infusion over 15 min.

.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women scheduled for an elective cesarean section with at least one risk factor for postpartum hemorrhage

Exclusion Criteria:

* suspected coagulopathy
* women refuse to participate
* emergent cesarean section
* allergy to misoprostol or tranexamic acid or carbetocin
* known deep venous thrombosis
* general anesthesia

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women scheduled for an elective cesarean section with at least one risk factor for postpartum hemorrhage
Enrollment: 400 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants require additional pharmacological uterotonic. | ist 24 hours post operative
  Number of participants need extra uterotonic

SECONDARY OUTCOMES:
intraoperative blood loss | during the operation
  amount of blood loss during cesarean section
post operative blood loss | 24 hours post operative
  amount of blood loss after cesarean section
Number of participants need for blood transfusion | 24 hours post operative
  Number of participants needed for transfusion

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No